CLINICAL TRIAL: NCT07252154
Title: Modified Technique for Nuclear Phacoemulsification in Brown Cataractous Nucleus
Brief Title: Modified Nuclear Phacoemulsification in Brown Cataract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hassan Lotfy Fahmy, Prof, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17209067
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Brown Cataract
Keywords: phaco; hard nucleus
MeSH Terms: interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Brown cataract (Experimental): doing phacoemulsification as usual, but we stop when the gutter becomes half the thickness of the nucleus, then we use the tip of the phaco as irrigation for 30 seconds. the nucleus will become softer
  Interventions: Procedure: phacoemulsification

INTERVENTIONS:
Procedure: phacoemulsification — doing phacoemulsification as usual but we stop when the gutter becomes half the thickness of the nucleus then we use tip of the phaco as irrigation for 30 seconds. the nucleus will become more softer

SUMMARY:
Irrigation of the nucleus with saline for 30 seconds after creating the central groove.

DETAILED DESCRIPTION:
The hard nucleus is physiologically immune against water flow from out to inside the nucleus but we discovered that it is not immune against the flow of water from inside the nucleus to outside. So, we are doing phacoemulsification as usual, but we stop when the gutter becomes half the thickness of the nucleus, then we use the tip of the phaco as irrigation for 30 seconds. the nucleus will become softer.

. As we know, the nucleus of the lens has the highest concentration of crystalline (high osmotic pressure), so the water will flow from the center of the nucleus to the outer surface without any resistance, and all adhesions and bonds between lens fibers will be broken at once, and the nucleus becomes softer.

ELIGIBILITY:
Inclusion Criteria:

* Brown cataract

Exclusion Criteria:

* white cataract
* soft cataract

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
phaco time | 60 seconds
  time of ultrasound power

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut univercity, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No